CLINICAL TRIAL: NCT03473522
Title: Effects of Transcranial Direct Current Stimulation Combined With Therapeutic Exercises in Patients With Parkinson's Disease: Randomized Clinical Trial
Brief Title: Effects of tDCS Combined With Therapeutic Exercises in Patients With Parkinson's Disease.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alessandra Tanuri Magalhães (Other)
Collaborators: Foundation for Research Support of the State of Piauí (Other)
Responsible Party: Sponsor-Investigator, Alessandra Tanuri Magalhães, Full Professor of Physical Therapy Department, Universidade Federal do Piauí
Organization: Universidade Federal do Piauí (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.085.438
Record Dates: First submitted 2018-02-07; First posted 2018-03-22 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
Keywords: Transcranial Direct Current Stimulation; therapeutic exercises; Parkinson
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation; Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, sham-controlled, clinical trial involving two types of intervention: (1) Physical therapy + active tDCS; (2) Physical therapy + sham tDCS.
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS +Exercise Therapy (Experimental): Anodal tDCS (2mA of intensity, for twenty minutes) over the motor cortex representation of trunk and lower limbs. Immediately after tDCS application all the patients will participate in an exercise therapy protocol involving balance control, strength,
  Interventions: Device: tDCS; Behavioral: Exercise Therapy
- Sham tDCS+ Exercise Therapy (Sham Comparator): Anodal tDCS (2mA of intensity, for twenty minutes but thirdy seconds ON) over the motor cortex representation of trunk and lower limbs.
  Interventions: Device: tDCS; Behavioral: Exercise Therapy

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation is a modulation technique of neuronal excitability which has very promising results in Parkinson's disease. In addition to the possibility of increasing the excitability of areas to tDCS, it can also facilitate the execution of the exercises by increasing the excitability of the primary motor cortex and changing the recruitment strategies of the motor units.
  Other Names: non invasive brain stimulation
Behavioral: Exercise Therapy — Therapeutic exercises will be based on the literature (O'Sullivan and Schmitz 2004, Klamroth et al 2016, Reynolds et al., 2016, Pérez et al 2016, Smania et al., 2010, Pastor et al., 1993, Traub et al., 1980, Schoneburg et al., 2013) Each session will be divided into warm-up exercises; balance and relaxation, with a duration of 50 minutes and a frequency of 3 times a week. Training progresses and intensifies every two weeks. The subjects will perform five repeated movements of each exercise, evolving according to the condition of each patient (according to the Hoehn and Yahr staging scale).
  Other Names: Physiotherapy

SUMMARY:
Parkinson's disease is a progressive, degenerative neurological disease associated with profound changes in the quality of life of its survivors. Therapeutic exercises are widely employed in the attempt to delay or minimize disease progression, characterized by significant motor and sensory deficits. Recent evidence has demonstrated the potential use of transcranial direct current stimulation (TDCs) as a complement to therapeutic exercises. However, few studies have investigated the effects of TDCs combined with therapeutic exercises in patients with Parkinson's disease. This study aims to investigate the effect of TDCs combined with therapeutic exercises in people with Parkinson's disease. Thirty patients will be randomized into two distinct groups to receive either TDCs(anodal) + therapeutic exercises or TDCs (sham) + therapeutic exercises for 24 sessions over a five-week period. The primary clinical outcome (balance) and secondary outcomes (functional capacity, quality of life and perception of overall effect) will be collected before treatment after two and five weeks at month 3 and month 6 after randomization. The data will be collected by a blind examiner to the treatment allocation.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo-controlled experimental design will be used. The 30 participants will be randomized into two groups: (1) TDCs(anodal) + therapeutic exercises and (2) TDCs (sham) + therapeutic exercises. The treatment will be performed for 8 weeks, with three sessions per week, totaling 24 sessions of electrostimulation and therapeutic exercises. The primary variable (balance), secondary outcomes and other outcomes will be assessed before and after treatment. Follow-up of patients will be conducted at 8, 12 and 24 weeks after randomization. All evaluations will be performed by a single researcher who, like the patients, will not know which stimulation group will be participating. Patients diagnosed with Parkinson's who seek treatment at the Clinical School of Physiotherapy of the Federal University of Piauí will receive detailed instructions on the present study. The physiotherapist responsible for evaluations will explain the objectives of the study, possible treatments, eligibility criteria and potential risks arising from the application of brain stimulation and therapeutic exercises. Patients who agree to the conditions and sign the consent form may participate in the study. Participants who meet the eligibility criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of idiopathic Parkinson's disease present for at least 12 months,
* spontaneous demand for treatment,
* in clinical follow-up and pharmacological treatment by a responsible physician,
* Parkinson's classification of 1.5-3 according to the Hoehn and Yahr scale,
* absence of cardiovascular diseases and musculoskeletal,
* signing of the free and informed consent form.

Exclusion Criteria:

* Use any associated orthopedic device to aid gait or balance control,
* signs of severe dementia (evaluated by the Mini-Mental State Examination - MMSE),
* diagnosis of other neurological disorders (including those of central and peripheral nature)
* previous treatment with tDCS,
* medical diagnosis of psychiatric illnesses with the use of centrally acting medications (depressants)
* the use of pacemakers or other implanted devices.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change From balance | 8 weeks after randomization
  Balance will be evaluated using a force plate to record center of pressure displacement (COP) in antero-posterior (AP) and Mediolateral (ML) axes in centimeters. Other variables such as area (cm²), speed AP and ML(cm/s), frequency (Hz) and Entropy (no unit) will be derived from COP displacement.

SECONDARY OUTCOMES:
Change From balance | 3 and 6 months after randomization
  Balance will be evaluated using a force plate to record center of pressure displacement (COP) in antero-posterior (AP) and Mediolateral (ML) axes in centimeters. Other variables such as area (cm²), speed AP and ML(cm/s), frequency (Hz) and Entropy (no unit) will be derived from COP displacement.
Change From Unified Parkinson´s Disease Rating Scale | 8 weeks, 3 and 6 months after randomization
  The Unified Parkinson's Disease Rating evaluate is composed of 42 questions, divided into 4 parts: motor symptoms; mental activity, behavior and mood; activities of daily living; complications of drug therapy. The mental activity, behavior and humor part counts of 4 questions being the score ranging from 0 to 4 totaling 16 points. The daily life activity part consists of 13 questions that range from 0 to 4 scores totaling 52 points. The motor symptoms part consists of 14 questions, in which some of them have to be applied independently for each member. Thus, there are 27 observations that vary the score from 0 to 4, totaling 108 points. Part of the complications of drug therapy consists of 23 questions in which 4 vary the score from 0 to 4 and 7 questions vary the score from 0 to 1 totaling 23 points. Thus, the scoring of this scale varies between 0 and 199 in that the higher the score the greater the impairment and the closer to zero the more tendency to normality
Change From Parkinson Disease Quality of Life | 8 weeks, 3 and 6 months after randomization
  Parkinson Disease Quality of Life is a questionnaire consists of 37 items, subdivided into four domains: parkinsonian symptoms (14 items), systemic symptoms (7 items), emotional function (7 items) social function (9 items). The score ranges from 1 (all time), 2 (almost always), 3 (sometimes), 4 (few times) and 5 (never). The score of each domain is determined by the average of the points of each domain. The sum of the average score of each domain is made and high scores refers to the individual's better perception regarding his or her quality of life.
Change in the perception scale of the overall effect | 8 weeks, 3 and 6 months after randomization
  Perception scale of the overall effect evaluates the level of perception of recovery of the patient in relation to the treatment comparing the beginning of the symptoms with the last days. It is a numerical scale of 11 points ranging from -5 to +5, being - 5: extremely worse; zero: no modification; and +5: fully recovered, with the highest score representing greater recovery
Maximal Isometric Voluntary Contraction | 8 weeks, 3 and 6 months after randomization
  Peak and average force (Kg or Newton) and time to peak (seconds) will be collected during the maximal Isometric contraction of knee extensor muscles.
Tampa Scale for Kinesiophobia (TSK) | 8 weeks, 3 and 6 months after randomization
  Irrational, and debilitating fear of movement and activity resulting from a feeling of vulnerability to painful injury or re-injury. Its a 17-item scale.

OTHER OUTCOMES:
Geriatric Depression Scale (GDS) | 8 weeks, 3 and 6 months after randomization
  Assessment of emotional function with GDS. Its a 15 item scale

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Piauí, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No